CLINICAL TRIAL: NCT02307019
Title: Intervention on Caregivers Caring for Patients Poststroke With Upper Limb Apraxia: Randomized Clinical Trial
Brief Title: Intervention on Caregivers Caring for Patients Poststroke With Upper Limb Apraxia
Acronym: CPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Encarnación Aguilar Ferrandiz, Intervention on caregivers caring for patients poststroke with upper limb apraxia: Randomized Clinical Trial, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Caregiver patients apraxia
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Performance Anxiety; Emotional Stress
Keywords: Caregivers; Apraxias; Stroke; Cerebral Stroke; Rehabilitation; Pragmatic Clinical Trials as Topic
MeSH Terms: conditions — Stress, Psychological; Apraxias; Stroke | interventions — Caregivers

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Program on specific prevention of health (Experimental): The caregivers will be randomly assigned to an experimental group, to receive the program on specific prevention of health. The workshop will be performed twice a month, two hours a day, during a 4-week period.
  Interventions: Other: Program on specific prevention of health
- Program on general prevention of health (Active Comparator): Control group will receive an intervention by mean of a general health program to manage the common situations when a caregiver is caring for a patient with dependency. The workshop will be performed two a month, two hours a day, during a 4-week period.
  Interventions: Other: Program on general prevention of health

INTERVENTIONS:
Other: Program on specific prevention of health — The intervention will be centered in provide effective tools to manage each situation presented while a caregiver cares for patients poststroke with upper limb apraxia. Moreover, the workshops will be focused on the balance between the assistance provided by the caregiver and the improvement and the increase the autonomy and independence of the patients. Finally, we will provide skills and strategies to the caregiver for enhancing the environment adaptation of the patients.
  Other Names: Program of specific intervention for caregivers
  Arms: Program on specific prevention of health
Other: Program on general prevention of health — The general health educative program will consist in an educational workshop for caregivers where they are taught the habitual guidelines to caring for patients in situation of dependency.
  Other Names: Program on traditional intervention for caregivers
  Arms: Program on general prevention of health

SUMMARY:
The purpose of this study is to analyze the effects of a intervention on a specific health prevention/intervention program aimed at caregivers of mild and moderate patients post stroke with upper limb apraxia in comparison to a control group with a no specific formation in that kind of patients.

DETAILED DESCRIPTION:
Patients with Upper limb apraxia after stroke have severe problems to adapt their daily life.

The upper limb apraxia syndrome affects the performance of skilled movements carried out by the upper limbs and provoke that many patients´activities have to be made by their main caregiver or carers.

Caregivers usually have to occupy much time and efforts for caring their familiar or client, and it can result in a overload in different areas of the caregiver health.

Few data are available on the effectiveness of interventions in caregivers that informally works with that kind of patients.

The specific prevention health program is based on improving the awareness of the assistance that the caregivers provide, and knowing the process of the information that carer has to give to the patient while the patients have their activities made.

ELIGIBILITY:
Inclusion Criteria:

* Having an habitual role of carer (informal or formal).
* Being caring a mild-moderate poststroke patient with upper limb apraxia.
* Subjective manifestations of overload in the role as carer.
* More than two month as carer.

Exclusion Criteria:

* Uncooperativeness
* Being formed in the care of that kind of patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Stroke Impact Scale (SIS-16) at 8 weeks | Eight weeks
Change from Baseline in Stroke Impact Scale (SIS-16) at 16 weeks | Sixteen weeks

SECONDARY OUTCOMES:
Change from Baseline in Barthel index at 8 weeks | Eight weeks
Change from Baseline in Barthel index at 16 weeks | Sixteen weeks
Change from Baseline in Disabilities of the Arm, Shoulder and Hand (Quick-DASH) at 8 weeks | Eight weeks
Change from Baseline in Disabilities of the Arm, Shoulder and Hand (Quick-DASH) at 16 weeks | Sixteen weeks
Change from Baseline in General health questionnaire (GHQ-28) at 8 weeks | Eight weeks
Change from Baseline in General health questionnaire (GHQ-28) at 16 weeks | Sixteen weeks
Change from Baseline in Zarit questionnaire at 8 weeks | Eight weeks
Change from Baseline in Zarit questionnaire at 16 weeks | Sixteen weeks
Change from Baseline in family APGAR at 8 weeks | Eight weeks
Change from Baseline in family APGAR at 16 weeks | sixteen weeks
Change from Baseline in Duke-UNC-11 questionnaire of functional social support at 8 weeks | Eight weeks
Change from Baseline in Duke-UNC-11 questionnaire of functional social support at 16 weeks | Sixteen weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mª Encarnacion ME Aguilar, PhD, Principal Investigator — Department of Physiotherapy. Faculty of Sciences of Health. University of Granada (Granada). Spain
Locations (1):
- University of Granada, Granada, Andalusia, Spain